CLINICAL TRIAL: NCT03382639
Title: A Phase 2, 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate Efficacy, Safety, Tolerability, and Pharmacokinetics of 3 Dose Levels of TAK-831 in Adjunctive Treatment of Adult Subjects With Negative Symptoms of Schizophrenia
Brief Title: A Study to Evaluate 3 Dose Levels of Luvadaxistat of Adults With Negative Symptoms of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TAK-831-2002; 2017-003471-54 (EudraCT Number); U1111-1201-2722 (Other: WHO)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Schizophrenia
Keywords: Drug therapy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Luvadaxistat 50 milligrams (mg) (Experimental): Participants received luvadaxistat 50 mg orally once daily (QD) for 12 weeks (Days 1 to 84).
  Interventions: Drug: Luvadaxistat
- Luvadaxistat 125 mg (Experimental): Participants received luvadaxistat 125 mg orally QD for 12 weeks (Days 1 to 84).
  Interventions: Drug: Luvadaxistat
- Luvadaxistat 500 mg (Experimental): Participants received luvadaxistat 500 mg orally QD for 12 weeks (Days 1 to 84).
  Interventions: Drug: Luvadaxistat
- Placebo (Placebo Comparator): Participants received placebo (matching luvadaxistat) orally QD for 12 weeks (Days 1 to 84).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Luvadaxistat — TAK-831 tablets.
  Other Names: TAK-831; NBI-1065844
  Arms: Luvadaxistat 125 mg; Luvadaxistat 50 milligrams (mg); Luvadaxistat 500 mg
Drug: Placebo — Luvadaxistat placebo-matching tablets.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether add-on luvadaxistat is superior to placebo on the Positive and Negative Syndrome Scale Negative Symptom Factor Score (PANSS NSFS).

DETAILED DESCRIPTION:
The drug being tested in this study is called luvadaxistat. Luvadaxistat is being tested to treat negative symptoms in participants who have schizophrenia.

Participants will be randomly assigned (by chance, like flipping a coin) to one of the four treatment groups in the double-blind period-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Luvadaxistat 50 mg once daily
* Luvadaxistat 125 mg once daily
* Luvadaxistat 500 mg once daily
* Placebo once daily

ELIGIBILITY:
Inclusion Criteria:

1. Has a current diagnosis of schizophrenia as defined by the Mini International Neuropsychiatric Interview (MINI) 7.0.2 for Psychotic Disorders for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and the general psychiatric evaluation.
2. Initial diagnosis must be greater than or equal to (>=1) year from screening.
3. Is receiving primary background antipsychotic therapy (other than clozapine) at a total daily dose between 2 and 6 mg of risperidone equivalents. Concomitant treatment with a sub-therapeutic dose of a second antipsychotic may be permitted with sponsor or designee approval if used to treat specific symptoms, such as insomnia or anxiety (for example, quetiapine 25-50 mg or its equivalent as needed for anxiety), but not if it is used for refractory positive psychosis symptoms.
4. Is treated with a stable regimen of psychotropic medications with no clinically meaningful change (no increase in dose, less than or equal to [<=] 25 percent [%] decrease in dose for tolerability) in the prescribed dose for 2 months before the screening visit and no dose adjustment is anticipated throughout study participation up to the Day 84/early termination visit.
5. Has a BNSS total score (12-item, excluding number 4) >=28; stable Single-blind Placebo Run-in and baseline BNSS total (12-item, excluding number 4) scores (<= 20% change from the screening score).
6. Has no more than moderate-severe (<=5) rating on PANSS positive symptom items P1, P3, P4, P5, P6, or unusual thought content (G9), with a maximum of 2 of these items rated '5'; no more than moderate (<=4) rating on conceptual disorganization (P2).
7. There is evidence that the participant has stable symptomatology >=3 months prior to the screening visit (example, no hospitalizations for schizophrenia, no emergency room admission due to symptoms of schizophrenia, no increase in level of psychiatric care due to worsening of symptoms of schizophrenia).
8. Have an adult informant who will be able to provide input for completing study rating scales, including the PANSS and SCoRS (for example, a family member, social worker, caseworker, residential facility staff, or nurse who spends >=4 hours/week with the participant) and is considered reliable by the investigator. The informant must be able and willing to provide written informed consent and to participate in at least 1 in-person interview, then be able to provide continuing input by attending each clinical assessment visit or via participating in a telephone interview for other study visits that include the PANSS or SCoRS endpoints.

Exclusion Criteria:

1. Has a lifetime diagnosis of schizoaffective disorder; a lifetime diagnosis of bipolar disorder; or a lifetime diagnosis of obsessive compulsive disorder based on the MINI combined with the general psychiatric evaluation.
2. Has a recent (within the last 6 months) occurrence of panic disorder, depressive episode, or other comorbid psychiatric conditions currently requiring clinical attention based on the MINI for DSM-5 and the general psychiatric evaluation.
3. Has a diagnosis of substance use disorder (with the exception of nicotine dependence) within the preceding 6 months based on the MINI for DSM-5 and the general psychiatric evaluation.
4. Is participating in a formal structured nonpharmacological psychosocial therapeutic treatment program (cognitive remediation, cognitive-behavioral therapy, intensive symptom/vocational rehabilitation) for a duration of less than (<) 3 months before randomization. In addition, initiation of such nonpharmacological treatment programs is not permitted during study participation through the Day 84 visit.
5. The participant exhibits more than a minimal level of antipsychotic-induced parkinsonism symptoms, as documented by a score on the modified Simpson Angus Scale (SAS) (excluding item number 10, Akathisia) greater than (>) 6.
6. Has evidence of depression as measured by a Calgary Depression Scale Score (CDSS) > 9.
7. Is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property, or the participant has attempted suicide within the past year prior to screening. Participants who have positive answers on item number 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) (based on the past year) prior to randomization are excluded.
8. Has a history of brain trauma associated with loss of consciousness for >15 minutes.
9. Diagnosis of schizophrenia occurred prior to 12 years of age.
10. Has received electroconvulsive therapy within 6 months (180 days) before Screening.
11. Has a history of developmental intellectual disability or mental retardation.
12. Antipsychotic plasma levels for the participant's primary background antipsychotic are below the minimum acceptable concentration criteria per the Antipsychotic Reference document at the screening or placebo run-in visits. This criterion is not applicable to participants on a primary background antipsychotic for which a clinical assay is unavailable.
13. Is treatment resistant. Treatment resistance is defined as prior nonresponse of positive symptoms of schizophrenia to 2 courses of treatment with antipsychotics of different chemical classes for at least 4 weeks, each at doses considered to be effective.
14. Does not have a stable residence or is homeless.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 256 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (16):
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Synergy Clinical Research Center, Lemon Grove, California
  - Semel Institute for Neuroscience and Human Behavior, Los Angeles, California
  - Excell Research, Oceanside, California
  - NRC Research Institute, Orange, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Connecticut Mental Health Center - Yale University, New Haven, Connecticut
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - The Dr. Alan & Diane Breier Prevention and Recovery Center for Early Psychosis, Indianapolis, Indiana
  - Center for Behavioral Health, LLC, Gaithersburg, Maryland
  - Cherry Health, Grand Rapids, Michigan
  - Manhattan Psychiatric Center, New York, New York
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Community Clinical Research, Inc., Austin, Texas
  - Core Clinical Research, Everett, Washington
- Bulgaria (7):
  - State Psychiatric Hospital - Lovech, Lovech
  - State Psychiatric Hospital "Sv. Ivan Rilski", Novi Iskar, Novi Iskar
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - Medical Centre "Sv. Naum", Sofia
  - DCC "Sv. Vrach and Sv. Sv. Kuzma and Damyan", OOD, Sofia
  - DCC "Mladost M" - Varna, OOD, Varna
  - Mental Health CenterVratsa EOOD, Vratsa
- Czechia (6):
  - Narodni ustav dusevniho zdravi, Klecany
  - A-SHINE s.r.o., Pilsen
  - CLINTRIAL s.r.o., Prague
  - PRAGTIS s.r.o., Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - MUDr. Simona Papezova s.r.o., Prague
- Germany (4):
  - Zentralinstitut fuer Seelische Gesundheit, Mannheim, Baden-Wurttemberg
  - Studienzentrum Nordwest, Westerstede, Lower Saxony
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
- Italy (5):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliera Universitaria- Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Poland (7):
  - Przychodnia Srodmiescie Sp. z o. o., Bydgoszcz
  - NZOZ Syntonia, Gdynia
  - Care Clinic, Katowice
  - NZOZ Poradnia Zdrowia Psychicznego, Kobierzyce
  - Centrum Medyczne Plejady, Krakow
  - Medycyna Milorzab, Lodz
  - Centrum Medyczne "Luxmed" Sp. z o.o., Lublin
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Ukraine (7):
  - Regional Psychoneurological Hospital #3, Ivano-Frankivsk
  - CIH Kharkiv Regional Clinical Psychiatric Hospital #3, Kharkiv
  - Kyiv CH on Railway Transport #2 of Branch Center of Healthcare Public Company Ukr Railway, Kyiv
  - CI Kirovograd RPH Male dept#11,Female dep#17 Donetsk NMU, Nove, Kropyvnytskiy
  - Ternopil RCCPH Depts of Psychiatry #2 (m) & Psychiatry #4 (f) Ternopil I.Ya. Gorbachevskyi SMU, Ternopil
  - Transcarpathian Regional Narcological Dispensary, Uzhhorod
  - Zhytomyr Regional Psychiatric Hospital #1, Zarichany Vil.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murthy V, Hanson E, DeMartinis N, Asgharnejad M, Dong C, Evans R, Ge T, Dunayevich E, Singh JB, Ratti E, Galderisi S. INTERACT: a randomized phase 2 study of the DAAO inhibitor luvadaxistat in adults with schizophrenia. Schizophr Res. 2024 Aug;270:249-257. doi: 10.1016/j.schres.2024.06.017. Epub 2024 Jun 28. PMID 38943928

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a screening period of up to 28 days, a 14-day single-blind placebo run-in period, a 12-week double-blind treatment period and a safety follow-up visit. Randomization was stratified by age at screening (<35 and ≥35 years). The allocation ratio was 2:2:2:3 to the 3 luvadaxistat groups and placebo group, respectively.
Groups:
- Placebo: Participants received placebo (matching luvadaxistat) orally once daily (QD) for 12 weeks (Days 1 to 84).
- Luvadaxistat 50 Milligrams (mg): Participants received luvadaxistat 50 mg orally QD for 12 weeks (Days 1 to 84).
Period: Overall Study
Arm/Group | Placebo | Luvadaxistat 50 Milligrams (mg) | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Started | 87 | 58 | 56 | 55
Completed | 76 | 53 | 52 | 47
Not Completed | 11 | 5 | 4 | 8
Not completed — Adverse Event | 2 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 2 | 3
Not completed — Unsatisfactory therapeutic response | 1 | 0 | 0 | 0
Not completed — Noncompliance with study drug during the DBTP | 1 | 2 | 1 | 1
Not completed — Other | 2 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) will included all participants who were randomized and received at least 1 dose of the study drug during the Double-Blind Treatment Period.
Groups:
- Luvadaxistat 50 mg: Participants received luvadaxistat 50 mg orally QD for 12 weeks (Days 1 to 84).
- Total: Total of all reporting groups
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg | Total
Number analyzed (Participants) | 87 | 58 | 56 | 55 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 87 | 58 | 56 | 55 | 256
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 22 | 22 | 88
  Male | 63 | 38 | 34 | 33 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 1 | 8
  Not Hispanic or Latino | 19 | 12 | 18 | 8 | 57
  Unknown or Not Reported | 65 | 44 | 36 | 46 | 191
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 0 | 3
  Asian | 2 | 0 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 5 | 5
  Black or African American | 10 | 9 | 9 | 0 | 28
  White | 70 | 46 | 42 | 50 | 208
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the PANSS NSFS at Week 12
Description: PANSS assesses the positive symptoms, negative symptoms and general psychopathology associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Here, the PANSS NSFS subscale consists of 7 items which assess the negative symptoms with subscale score ranging from 7 to 49, where a higher score indicates greater severity. Baseline was defined as the last observed value before the first dose of study treatment. Results are reported as least squares (LS) mean change from baseline at Week 12, determined using a mixed model for repeated measures (MMRM). A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: The FAS included all randomized participants who received at least 1 dose of double-blind study treatment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 87 | 58 | 56 | 55
scores on a scale | -3.1 (0.44) | -3.3 (0.52) | -3.4 (0.51) | -2.5 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Luvadaxistat 50 mg; Test type: Superiority; p = 0.426, Mixed Models Analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-1.4 to 1.2], Standard Error of Mean 0.66
Statistical Analysis 2: Comparison: Placebo vs Luvadaxistat 125 mg; Test type: Superiority; p = 0.725, Mixed Models Analysis; LS Mean Difference = -0.2, 95% CI 2-sided [-1.5 to 1.1], Standard Error of Mean 0.66
Statistical Analysis 3: Comparison: Placebo vs Luvadaxistat 500 mg; Test type: Superiority; p = 0.808, Mixed Models Analysis; LS Mean Difference = 0.6, 95% CI 2-sided [-0.7 to 1.9], Standard Error of Mean 0.68

2. Secondary Outcome: Change From Baseline on the PANSS NSFS at Week 4 and Week 8
Description: PANSS assesses the positive symptoms, negative symptoms and general psychopathology associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Here, the PANSS NSFS subscale consists of 7 items which assess the negative symptoms with subscale score ranging from 7 to 49, where a higher score indicates greater severity. Baseline was defined as the last observed value before the first dose of study treatment. Results are reported as LS mean change from baseline at Weeks 4 and 8, determined using a MMRM. A negative change from baseline indicates improvement.
Time Frame: Baseline and Weeks 4 and 8
Population: The FAS included all randomized participants who received at least 1 dose of double-blind study treatment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 87 | 58 | 56 | 55
scores on a scale
  Change at Week 4 | -1.7 (0.32) | -1.6 (0.39) | -1.8 (0.38) | -1.4 (0.40)
  Change at Week 8 | -2.8 (0.39) | -2.2 (0.46) | -2.6 (0.45) | -2.3 (0.49)

3. Secondary Outcome: Change From Baseline on the Brief Negative Symptom Scale (BNSS) Total Score (12-item) at Week 12
Description: The BNSS is a 13-item instrument that measures 5 domains of negative symptoms: blunted affect, alogia, asociality, anhedonia and avolition. All items in the BNSS are rated on a 7-point (0-6) scale, with anchor points generally ranging from symptoms being absent (0) to severe (6). Here, the BNSS total score (12-item, excluding item 4) was calculated by summing the 12 individual items; total score range of 0 to 72, where a higher score indicates higher severity of negative symptoms. Participants required a BNSS total score ≥28 to be eligible for the study (excluding item 4). Baseline was defined as the last observed value before the first dose of study treatment. Results are reported as LS mean change from baseline at Week 12, determined using a MMRM. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: The FAS included all randomized participants who received at least 1 dose of double-blind study treatment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 87 | 58 | 56 | 55
scores on a scale | -7.1 (1.04) | -8.9 (1.22) | -8.0 (1.22) | -6.0 (1.30)

4. Secondary Outcome: Change From Baseline on the Brief Assessment of Cognition in Schizophrenia (BACS) Composite Score at Week 12
Description: BACS is a cognition assessment battery and includes brief assessments of reasoning and problem solving, verbal fluency, attention, verbal memory, working memory and motor speed. The primary measure from each test is standardized by creating T-scores whereby the mean of the test session of a healthy person is set to 50 and the standard deviation set to 10. A composite T-score is calculated by averaging the 6 standardized primary measures. The composite T-score indicates how much higher or lower the participants cognition is compared to a healthy person. Lower T-scores are indicative of lower cognitive performance. Baseline was defined as the last observed value before the first dose of study treatment. Results are reported as LS mean change from baseline at Day 12, determined using a MMRM.
Time Frame: Baseline and Week 12
Population: The FAS included all randomized participants who received at least 1 dose of double-blind study treatment.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 87 | 58 | 56 | 55
T-score | 2.3 (0.83) | 4.6 (0.97) | 3.5 (0.96) | 2.3 (1.04)

5. Secondary Outcome: Change From Baseline on the Clinical Global Impression-Schizophrenia Severity (CGI-SCH-S) Negative Symptoms Score at Week 12
Description: The CGI-SCH scale is an adapted version of the CGI scale that is designed to assess global illness status in participants with schizophrenia. CGI-SCH-S is a 7-point scale that requires the investigator to rate the severity of the participant's illness at the time of assessment. Here, CGI-SCH-S negative symptoms score assesses the severity of illness for negative symptoms on the following 7-point scale: 1. normal, not at all ill; 2. borderline mentally ill; 3. mildly ill; 4. moderately ill; 5. markedly ill; 6. severely ill; or 7. among the most extremely ill. Baseline was defined as the last observed value before the first dose of study treatment. The number of participants with each CGI-SCH-S negative symptoms score at baseline and at Week 12 is reported.
Time Frame: Baseline and Week 12
Population: The FAS included all randomized participants who received at least 1 dose of double-blind study treatment. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 71 | 51 | 49 | 45
Participants
  Baseline: Normal, not at all ill (1) | 0 | 0 | 0 | 0
  Baseline: Borderline mentally ill (2) | 0 | 0 | 1 | 0
  Baseline: Mildly ill (3) | 3 | 3 | 1 | 3
  Baseline: Moderately ill (4) | 36 | 28 | 25 | 22
  Baseline: Markedly ill (5) | 26 | 18 | 20 | 18
  Baseline: Severely ill (6) | 6 | 2 | 2 | 2
  Baseline: Among the most extremely ill (7) | 0 | 0 | 0 | 0
  Week 12: Normal, not at all ill (1) | 0 | 0 | 0 | 0
  Week 12: Borderline mentally ill (2) | 1 | 3 | 2 | 3
  Week 12: Mildly ill (3) | 13 | 14 | 12 | 11
  Week 12: Moderately ill (4) | 34 | 22 | 21 | 18
  Week 12: Markedly ill (5) | 20 | 11 | 13 | 12
  Week 12: Severely ill (6) | 3 | 1 | 1 | 1
  Week 12: Among the most extremely ill (7) | 0 | 0 | 0 | 0

6. Secondary Outcome: Clinical Global Impression Schizophrenia Improvement (CGI-SCH-I) Negative Symptoms Score at Week 12
Description: The CGI-SCH-I assesses the participant's improvement (or worsening). CGI-SCH-I requires the investigator to assess the participant's condition relative to baseline on a 7-point scale. Here, CGI-SCH-I negative symptoms score assesses the improvement for negative symptoms on the following scale: very much improved; 2. much improved; 3. minimally improved; 4. no change; 5. minimally worse; 6. much worse; or 7. very much worse. Baseline was defined as the last observed value before the first dose of study treatment. The number of participants with each CGI-SCH-I negative symptoms score at Week 12 is reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 71 | 51 | 49 | 45
Participants
  1 - Very much improved | 0 | 0 | 0 | 0
  2 - Much improved | 10 | 13 | 12 | 5
  3 - Minimally improved | 29 | 19 | 19 | 21
  4 - No change | 32 | 19 | 16 | 18
  5 - Minimally worse | 0 | 0 | 2 | 1
  6 - Much worse | 0 | 0 | 0 | 0
  7 - Very much worse | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline on the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Total Score at Week 12
Description: The SCoRS is an interview-based measure of cognitive functioning that is developed to specifically assess aspects of cognitive functioning in participants with schizophrenia. The items assess the 7 cognitive domains of attention, memory, reasoning and problem solving, working memory, processing speed, language functions and social cognition. The SCoRS total score is the sum of the 20 items and varies from 20 to 80 with 20 being the best outcome and 80 being the worst. Baseline was defined as the last observed value before the first dose of study treatment. Results are reported as LS mean change from baseline at Week 12, determined using a MMRM.
Time Frame: Baseline and Week 12
Population: The FAS included all randomized participants who received at least 1 dose of double-blind study treatment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 87 | 58 | 56 | 55
scores on a scale | -1.6 (0.66) | -3.8 (0.77) | -2.3 (0.77) | -1.8 (0.83)

8. Secondary Outcome: Change From Baseline on the PANSS Total Score at Week 12
Description: PANSS assesses the positive symptoms, negative symptoms and general psychopathology associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210, where a higher score indicates greater severity. Baseline was defined as the last observed value before the first dose of study treatment. Results are reported as LS mean change from baseline at Week 12, determined using a MMRM. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: The FAS included all randomized participants who received at least 1 dose of double-blind study treatment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 87 | 58 | 56 | 55
scores on a scale | -6.2 (1.00) | -7.2 (1.19) | -6.8 (1.18) | -5.0 (1.26)

9. Secondary Outcome: Change From Baseline on the PANSS Positive Symptom Factor Score (PSFS) at Week 12
Description: PANSS assesses the positive symptoms, negative symptoms and general psychopathology associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Here, the PANSS PSFS subscale consists of 7 items which assess the positive symptoms with subscale score ranging from 7 to 49, where a higher score indicates greater severity. Baseline was defined as the last observed value before the first dose of study treatment. Results are reported as LS mean change from baseline at Week 12, determined using a MMRM. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: The FAS included all randomized participants who received at least 1 dose of double-blind study treatment.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 87 | 58 | 56 | 55
scores on a scale | -0.8 (0.33) | -1.3 (0.39) | -1.3 (0.39) | -0.6 (0.42)

10. Secondary Outcome: Luvadaxistat Plasma Concentrations
Description: Blood samples were collected at pre-specified timepoints and plasma concentrations of luvadaxistat were measured. At Week 4, assessments were categorized as pre-dose or post-dose according to actual sampling time. Due to this, some participants may have had more than 1 record summarized for Week 4 pre-dose or Week 4 post-dose. Mean concentration on each visit was averaged from the observations over the time span of 24 hours post-dose or pre-dose.
Time Frame: Pre-dose on Day 1 and Week 4 and post-dose on Weeks 4, 6, 8 and 12
Population: PK analysis set included all randomized participants who received at least 1 dose of double blind study treatment and who had any available luvadaxistat plasma concentration data. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms / milliliter
Arm/Group | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 58 | 56 | 55
nanograms / milliliter
  Day 1 - Pre-dose: number analyzed (Participants) | 56 | 55 | 53
  Day 1 - Pre-dose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Week 4 - Pre-dose: number analyzed (Participants) | 45 | 31 | 42
  Week 4 - Pre-dose | 22.5 (44.44) | 106.5 (197.61) | 345.2 (653.08)
  Week 4 - Post-dose: number analyzed (Participants) | 58 | 56 | 53
  Week 4 - Post-dose | 79.0 (115.75) | 229.8 (368.27) | 480.2 (717.15)
  Week 6: number analyzed (Participants) | 55 | 53 | 47
  Week 6 | 83.60 (123.38) | 183.60 (257.44) | 409.3 (502.26)
  Week 8: number analyzed (Participants) | 54 | 53 | 46
  Week 8 | 109.3 (144.76) | 202.1 (294.60) | 366.80 (473.74)
  Week 12: number analyzed (Participants) | 51 | 48 | 44
  Week 12 | 61.50 (113.94) | 185.62 (258.73) | 356.0 (461.42)

ADVERSE EVENTS:
Time Frame: 12-week double-blind treatment period and up to 30 days follow-up: Day 1 up to Day 114.
Description: Treatment-emergent adverse events were defined as adverse events that occurred after the first dose of double-blind study treatment and up to 30 days after the last dose or early termination. The safety analysis set included all participants who were randomized and received at least 1 dose of double-blind study treatment.
Arm/Group | Placebo | Luvadaxistat 50 mg | Luvadaxistat 125 mg | Luvadaxistat 500 mg
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/58 | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 4/87 | 0/58 | 1/56 | 0/55
Other Adverse Events (participants affected / at risk) | 4/87 | 0/58 | 5/56 | 2/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=87) | Luvadaxistat 50 mg (N=58) | Luvadaxistat 125 mg (N=56) | Luvadaxistat 500 mg (N=55)
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=87) | Luvadaxistat 50 mg (N=58) | Luvadaxistat 125 mg (N=56) | Luvadaxistat 500 mg (N=55)
Headache (Nervous system disorders) | 4 | 0 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT03382639/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03382639/SAP_001.pdf